CLINICAL TRIAL: NCT05238662
Title: A Novel Technique for Degenerative Lumber Spine Fusion: Unilateral Pedicular Screws Fixation Combined With Contralateral Interbody Cage Fusion
Brief Title: Novel Technique Lumber Spine Fusion: Unilateral Pedicular Screws Fixation Combined With Contralateral Interbody Cage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, wael Abdelrahman Elmesallamy, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9181
Record Dates: First submitted 2022-02-07; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): pedicle screw fixation on one side and intervertebral cage on the other sided
  Interventions: Procedure: pedicle screw fixation on one side and intervertebral cage on the other sided
- Group B (Active Comparator): pedicle screw fixation and interbody cage on the same side
  Interventions: Procedure: pedicle screw fixation and interbody cage on the same side

INTERVENTIONS:
Procedure: pedicle screw fixation on one side and intervertebral cage on the other sided — pedicle screw fixation on one side and intervertebral cage on the other sided
  Arms: Group A
Procedure: pedicle screw fixation and interbody cage on the same side — pedicle screw fixation and interbody cage on the same side
  Arms: Group B

SUMMARY:
● Null hypothesis (H0): Unilateral pedicle screw with contralateral interbody cage has better outcomes than unilateral pedicle screw fixation with ipsilateral cage.

● Alternative hypothesis (H1):

Unilateral pedicle screw with contralateral interbody cage gives the same outcomes as unilateral pedicle screw fixation with ipsilateral cage.

DETAILED DESCRIPTION:
Lumber interbody fusion is one of the commonest neurosurgical procedures. A lot of studies showed the value of unilateral approach which resulted in less cost, time and radiation exposure when use interbody cage with ipsilateral pedicular screws fixation in comparison to bilateral approach when use interbody cage with bilateral pedicular screws fixation.

Fusion rate, cage migration, and biomechanical stress were the main draw backs of unilateral approach by lumber interbody fusion with ipsilateral cage and screws. Cage size and location seemingly the main reasons with advice to use large cage and cage insertion in oblique fashion to cross the midline. This study was designed to solve these issues.

Sample size:

The Study will include 40 patients divided into two groups, each group containing 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Both sexes.
* Age (21-60) years old.
* Patients with monosegmental lumber degenerative spinal diseases including lumbar spondylosis, spondylolysis, spondylolisthesis grade one, or lumbar disc prolapse.

Exclusion Criteria:

* Patient refusal.
* Altered mental status.
* Patients with associated comorbidity interfere with surgery.
* Extremes of age.
* Multiple level lumbar degenerative disease
* Trauma
* Spinal tumour
* Active infection
* Previous lumbar operation

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of fusion status | up to 3 months
  Evaluation of fusion status using CT scan and Xray

SECONDARY OUTCOMES:
Back Pain | At 24 hours, 2 weeks and 3 months after surgery
  use of Visual Analogue Scale (VAS) as a 10-cm line labeled with (0= no pain and 10=worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Wael Elmesallamy, M.D, Principal Investigator — Zagazig University, Faculty of human medicine